CLINICAL TRIAL: NCT05426629
Title: The Use of Hydradermabrasion in the Scalp to Improve Scalp Health and Improve Outcomes in Androgenetic Alopecia
Brief Title: Hydraderm for Androgenic Alopecia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: IRB closed
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DERM-2021-30436
Record Dates: First submitted 2022-03-29; First posted 2022-06-22 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Androgenic Alopecia
Keywords: alopecia; hair loss; pattern hair loss; hydradermabrasion; female pattern hair loss; male pattern hair loss; dermatology
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Intervention Model Description: Every participant will receive the same treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): 4 sessions of treatment at 1-week interval for first 4 weeks 3 sessions of treatment each 4 weeks apart, at week 8, week 12 and week 16
  1 Follow-up visit: Follow up 4 weeks after the last treatment at week 20
  Interventions: Device: Venus Glow

INTERVENTIONS:
Device: Venus Glow — The Venus Glow hydradermabrasion device is a class 1 device trimodality dermal system consisting of vacuum, 360 degrees rotating tip and two jet streams of saline.
  Adjustable vacuum deep cleanses the pores by pulling up daily dirt and debris, dry and dead skin cells, and excess sebum from the stratum corneum. It helps increase the microcirculation.
  The 360-degree rotation helps in spreading the saline evenly, which is expelled from two ultra-fine jet streams. This micro massaging helps in faster release of nutrients from the skin. The jet stream is smaller than the average pore size measuring 50- 70 microns each, enabling the jet stream to deep clean each pore.

SUMMARY:
The study will be focused on evaluating the use of hydradermabrasion on the scalp. The study aims to assess the effect of this treatment on scalp health and hair growth.

ELIGIBILITY:
Inclusion Criteria:

* Participants who can give voluntary, written informed consent to participate in this study and from whom consent has been obtained including HIPAA Authorization
* Participants who have androgenetic alopecia
* Healthy men and women, ages 18 - 65 years of age
* Participants who understand the study and can follow study instructions and are willing to attend the required study visits
* Participants who agree to be photographed for research purposes and their identity may not be concealed in these photographs.
* Participants who agree to continue their same treatment they are on at the baseline visit for androgenetic alopecia, for the entire duration of the study without plans to stop, change or add additional treatments.
* Participants who agree to use the same shampoo for the duration of the study

Exclusion Criteria:

* Participants who have not had a change to hair loss treatment for 4 months prior to study enrollment
* Participants who have an active or known skin inflammation or infection within the treatment area.
* Participants who have an active or known acute skin allergies
* Participants who have any other scalp conditions including eczema, psoriasis, infection, or scars within the treatment area
* Participants of child-bearing potential who are not using an approved method of birth control (oral contraceptives, IUD, contraceptive implant, barrier methods with spermicide or abstinence). Females of non-childbearing potential are defined as post-menopausal (absence of menstrual bleeding for one year), hysterectomy, or bilateral oophorectomy.
* Participants who are pregnant, planning to become pregnant or breastfeeding. A urine pregnancy test will be done to rule out pregnancy.
* Immunosuppression
* Participants who are HIV+ / Hepatitis B + / Hepatitis C+
* Participants who have been diagnosed or have a known history of any hematopathology disorders
* Participants who have been diagnosed or have a known history of haemostasis disorders
* Participants who have been diagnosed or have a known history of an autoimmune diseases
* Participants who are undergoing chemotherapy
* Participants with a history of any skin cancer on the scalp
* Participants who have had skin biopsy or procedure on scalp in last month
* Participants who have an implantable devices such as a deep brain stimulator in or other implantable device on or near treatment area
* Non-English speakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-04-21 (Estimated); Study Completion 2025-04-21 (Estimated)

PRIMARY OUTCOMES:
Scalp Health- Erythema | Assessed at Visit 8
  Primary endpoints will be changes in the Erythema score from baseline to Visit 8. Erythema score is a scale from 0 to 4.
Scalp Health- ASFS | Assessed at Visit 8
  Primary endpoints will be changes in the Adherent Scalp Flaking Score (ASFS) from baseline to Visit 8. ASFS is a scale 0 to 10.
Scalp Health- Folliculitis | Assessed at Visit 8
  Primary endpoints will be changes in the folliculitis score from baseline to Visit 8. Foliculitis score is a scale from 0 to 3.
Hair Changes | Assessed at Visit 8
  HairMetrix scale evaluates degree of improvement hair density, total hair count per sq cm and patient sensory assessment of scalp and hair from baseline to after each treatment and the follow up visit. The global assessment scales are a scale from 0 to 3.

CONTACTS AND LOCATIONS:
Overall Officials: Ronda Farah, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No